CLINICAL TRIAL: NCT03933345
Title: Overdose Risk Management and Compensation in the Era of Naloxone
Brief Title: Overdose Risk Management and Naloxone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: Brandeis University (Other); Drexel University (Other); New York University (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Alexander Bennett, Principal Investigator and Deputy Director, National Development and Research Institutes, Inc.
Other Study IDs: 660
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Opioid Use
Keywords: Overdose Risk Behaviors; Opioids; Naloxone; Overdose
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who use illicit opioids: The study will recruit an adult-age (18+) sample of 600 people who use illicit opioids (either heroin or prescription opioid analgesics without a doctor's prescription) in New York City using Respondent Driven Sampling.
  Interventions: Other: Study provides naloxone to participants who wish to have it. Not required to accept naloxone and no control.

INTERVENTIONS:
Other: Study provides naloxone to participants who wish to have it. Not required to accept naloxone and no control. — At enrollment, participants will complete a detailed survey instrument establishing histories of substance use, naloxone exposure, and other potential barriers to the uptake of naloxone training. Because extant research establishes a clear public health and ethical imperative to provide PWUIO with naloxone, we will also offer all participants training to become naloxone-equipped OD responders at enrollment. We will follow the sample for two years using a mixed-methods approach involving text-message-based exposure tracking, monthly surveys using a state-of-the-art online data collection portal, and a qualitative subsample to ensure that naloxone exposures and changes in OD risk behavior are carefully tracked and contextualized by ethnographic data about the psychosocial and sociocultural mechanisms underlying participant experiences.

SUMMARY:
A growing body of research underscores the life- and cost-saving advantages of equipping people who use opioids with naloxone, but very little is known about: 1) barriers to naloxone awareness and access, and 2) the potential psychosocial and behavioral impacts of being "protected" by naloxone while engaging in overdose risk behaviors, of using naloxone on someone else, and of surviving an overdose in which naloxone is used. This research will provide insight into both of these domains to yield a richly contextualized understanding of the processes and mechanisms underlying changes in overdose risk behaviors related to naloxone access and use and will illuminate the disparities that may limit access to naloxone for some or result in compensatory behavior following naloxone exposure for others. Findings from this study will provide an empirical basis to strengthen and refine existing overdose prevention efforts and to design tailored interventions to engage opioid users who have recently survived or reversed an overdose.

DETAILED DESCRIPTION:
Drug overdose (OD) deaths in the United States nearly tripled between 1999 and 2014. During 2015 more than 50,000 people died from overdose nationwide, and almost two thirds (63.1%) involved opioids.1 In response, the number of opioid OD prevention programs offering naloxone has ballooned.2 Many states have sought to expand access through provision of the medication to EMT and police first-responders, over-the-counter availability at pharmacies, and emergency legislation providing for lay prescribing, largely within the context of opioid OD prevention programs serving people who use heroin or diverted prescription opioids (henceforth, people who use illicit opioids; PWUIO). As naloxone has become more commonplace, however, OD rates have continued to rise, and critical viewpoints about the failure of OD reversal efforts to deter subsequent high-risk behavior have begun to emerge from police,3 firefighers,4 EMS personnel,5 and news media,6-8 especially following the recent loss of pop-artist, Prince, to an opioid OD only days after being administered naloxone in an Illinois hospital.9 This study is responsive to a recent NIDA and FDA mandate for foundational naloxone research among active users of illicit opioids.10 Specifically, it assesses two main concerns at the heart of current policymaking related to opioid OD and naloxone. 1) Disparities in access to naloxone and obstacles to a willingness to be trained as a naloxone-carrying OD responder: Despite the critically important role PWUIO can play as OD responders,11-15 questions remain about differential awareness of and access to naloxone and OD response training among PWUIO. Even in NYC where city and state departments of health have led concerted and well-funded efforts to saturate the city with naloxone and OD reversal training, considerable limitations in coverage and training uptake still exist.16 Findings from our ongoing study of opioid OD risks among military veterans in NYC indicate that many PWUIO are still naloxone-naïve and, even after learning about its lifesaving utility, still decline no-cost naloxone and OD response training. 2) The poorly understood impacts of possessing naloxone, using naloxone on someone else, or having it used on oneself on PWUIO's subsequent OD rates and risk behaviors: An increasing number of studies seek to track the uses to which naloxone kits are put, but the broader behavioral impacts of exposure to naloxone on actual opioid-related risk behaviors have seen almost no empirical investigation since 2003 when a study of street-recruited PWUIO in San Francisco reported that 35% indicated that they intended to use more heroin than usual after receiving naloxone.17 Building on our current studies of naloxone use and related attitudes among opioid-using military veterans and other drug users we propose to recruit 600 adult-age (18+) people who use illicit opioids (i.e., heroin and/or diverted pharmaceutical opioids) in New York City using Respondent Driven Sampling. At enrollment, participants will complete a detailed survey instrument establishing histories of substance use, naloxone exposure, and other potential barriers to the uptake of naloxone training. Because extant research establishes a clear public health and ethical imperative to provide PWUIO with naloxone, we will also offer all participants training to become naloxone-equipped OD responders at enrollment. We will follow the sample for two years using a mixed-methods approach involving text-message-based exposure tracking, monthly surveys using a state-of-the-art online data collection portal, and a qualitative subsample to ensure that naloxone exposures and changes in OD risk behavior are carefully tracked and contextualized by ethnographic data about the psychosocial and sociocultural mechanisms underlying participant experiences.

Aim A - Describe factors associated with: 1) lifetime history of access to and use of naloxone and 2) uptake of no-cost naloxone and OD response training. We will test the following hypotheses:

HypA1 - Naloxone knowledge and exposure history will vary at enrollment, potentially revealing disparities based on background factors (e.g., SES, ethnicity, age, neighborhood) and individual level factors (e.g., mental health diagnoses, opioid use disorder severity, duration of opioid use) HypA2 - Interest in OD response training and naloxone at baseline will vary by background and individual-level factors.

Aim B - Describe longitudinal relationships between naloxone exposure (access to and use of naloxone) and overdose risk behaviors. We will test the following hypothesis:

HypB1 - Naloxone access and use exposures will have measurable impacts on opioid OD-related risk behaviors over time, potentially varying in degree and direction across subgroups of PWUIO.

Aim C (Qualitative) - Explore barriers to naloxone uptake and any identified secondary impacts (e.g., compensatory risk taking, positive change after a naloxone exposure such as risk reduction or treatment-seeking) in terms of opioid users' own experiences and perceptions.

By employing a longitudinal and mixed-methods design capable of detecting naloxone exposure impacts and also illuminating the various mechanisms that may undergird them in participants' own terms, this project holds serious policy and direct service implications for the refinement of naloxone training programs and OD risk interventions that target PWUIO. This research also holds the potential to identify varying naloxone impacts among PWUIO of different social and behavioral groups-such as people who inject drugs (PWID) vs. prescription opioid misusers, older vs. younger (or shorter- vs. longer-term) PWUIO, and male vs. female users-and can inform future efforts to tailor prevention and education to these distinct subpopulations.

ELIGIBILITY:
Inclusion criteria:

* Adult-age (18+)
* Current illicit opioid use (verified by rapid urine screen)
* Speak English
* Willing to participate

Exclusion Criteria:

• Unable to comprehend informed consent and/or study procedures.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will consist of 600 people who use illicit opioids in New York City.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Naloxone access | Lifetime (at baseline)
  Number of times offered naloxone
Naloxone uptake | Lifetime (at baseline)
  Number of times accepted naloxone when offered
Naloxone use | Lifetime (at baseline)
  Number of times used naloxone
Naloxone access | 24 months
  Number of times offered naloxone
Naloxone use | 24 months
  Number of times used naloxone
Overdose risk behaviors | 24 months
  Overdose Risk Behavior Scale - a 22 item validated scale that measures past 30-day overdose risk behaviors. See (Development of an Overdose Risk Behavioral Scale: ORBS; Pouget et al., 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenblum, Study Director — National Development & Research Institutes (NDRI)
Locations (2):
- United States (2):
  - 270 West 25th Street, New York, New York
  - National Development and Research Institutes, Inc., New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pouget ER, Bennett AS, Elliott L, Wolfson-Stofko B, Almenana R, Britton PC, Rosenblum A. Development of an opioid-related Overdose Risk Behavior Scale (ORBS). Subst Abus. 2017 Jul-Sep;38(3):239-244. doi: 10.1080/08897077.2017.1282914. Epub 2017 Jan 23. PMID 28113004